CLINICAL TRIAL: NCT04937842
Title: Efficacy and Safety of Radiotherapy or Chemotherapy Combined With Microtransplantation in the Treatment of Advanced and Relapsed Solid Tumors
Brief Title: Microtransplantation for Advanced and Relapsed Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Principal Investigator, dayong, director, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MST-ST-01
Record Dates: First submitted 2021-05-30; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Solid Tumors
Keywords: microtransplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MST (Experimental): standard chemotherapy with microtransplantation
  Interventions: Biological: microtransplantation, HLA-mismatched donor peripheral stem cell infusion
- CT (No Intervention): standard chemotherapy only, without microtransplantation

INTERVENTIONS:
Biological: microtransplantation, HLA-mismatched donor peripheral stem cell infusion — infusion of granulocyte colony stimulating factor (G-CSF) mobilized HLA-mismatched peripheral blood stem cells (GPBSC)
  Other Names: DSI
  Arms: MST

SUMMARY:
In this study, we will apply micro transplantation to the field of solid tumors to study the efficacy and safety of radiotherapy and chemotherapy combined with micro transplantation in the treatment of advanced / relapsed solid tumors.

DETAILED DESCRIPTION:
The eligible patients are assigned to the experimental group (microtransplantation group, MST group) or the control group (CT) according to the availability of suitable donors. In MST group, peripheral blood hematopoietic stem cells from HLA mismatched donors mobilized with granulocyte colony stimulating factor are infused after conventional chemotherapy and/or radiotherapy ; The CT group only received conventional chemotherapy and/or radiotherapy. According to the patient's past medical history, current tumor assessment results, and the latest cancer treatment guidelines, the individualized chemotherapy and / or radiotherapy plan for the patient is formulated after discussion by more than 3 oncologists. After each course of treatment, the efficacy and safety are evaluated. For the patients who are evaluated to be effective or stable (SD) after the first treatment, the second treatment of the same scheme will be given. Those who reach the disease control level will continue to be treated for 4 courses, with an interval of 28 days. The patients who failed to achieve the improvement of SD after two cycles of chemotherapy will be withdrawn from the study. Patients are allowed to receive any treatment, including symptomatic support treatment, after the end of treatment or withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients are 18-80 years old, regardless of gender or race;
* Advanced / relapsed solid tumors (small cell lung cancer, ovarian cancer, cervical cancer, gastric and colorectal cancer, sarcoma, head and neck tumor, etc.) are confirmed by clinical or histopathological diagnosis;
* More than two kinds of tumors are allowed;
* Karnofsky score ≥ 60, ECoG physical status ≤ 2;
* Sensitive to chemotherapy or radiotherapy;
* There are measurable lesions;
* There are suitable hematopoietic stem cell donors

Exclusion Criteria:

* have no suitable donor or donor refused
* patient refused to accept donor cells

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | 1 month
  Treatment related mortality
time of hematopoietic recovery | 1 month
  Absolute neutrophil count >500/mcL; Platelets ≥20,000/mcL

SECONDARY OUTCOMES:
overall response rate | 1year
  (markedly effective + effective) / number of patients × 100%

CONTACTS AND LOCATIONS:
Overall Officials: Yong Da, Principal Investigator — Department of Medical Oncology, Beijing Fengtai You'anmen Hospital
Locations (1):
- Beijing Fengtai You'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No